CLINICAL TRIAL: NCT00005335
Title: Genetic Epidemiology of Lipoprotein-Lipid Levels
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4192; R01HL044672 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis

SUMMARY:
To determine the contribution of polymorphic variation in candidate genes involved in lipid metabolism in determining quantitative lipoprotein-lipid levels and cardiovascular risk factors in Anglo and Hispanic populations of the San Luis Valley in southern Colorado. The candidate genes included those for A-IV, B, D, E, H, APO(a), LDL receptor, hepatic lipase, lipoprotein lipase, lethicin cholesterol acyletransferase (LCAT), and cholesteryl ester transfer protein.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Beginning in 1991, genetic variations in the gene products of A-IV, E, H, and APO(a) were determined by isoelectric focusing and SDS/immunoblotting; gene variations at the APOB, D, LDL receptor, hepatic lipase, lipoprotein lipase, and cholesteryl ester transfer protein were assayed by polymerase chain reaction protocols and by using cloned cDNA probes for restriction fragment length polymorphism (RFLP) analyses. Direct haplotype analyses of individuals employed a strategy using RFLP analysis combined with the use of allele specific oligonucleotides. Quantitative levels of apolipoprotein B, E, H and APO (a) were determined by immunological techniques. These data and prior data on levels of triglycerides, total cholesterol, HDL-, LDL- and HDL subfraction cholesterol were used in the quantitative genetic analysis. Estimates of the effect of alleles at each of the genetic loci on the quantitative apolipoprotein and lipoprotein levels employed the measured genotype approach. The effects of multisite haplotypes for RFLPs at various loci were estimated using the same methods. For common alleles in each system, estimates were made of the interaction of alleles at independent genetic loci in determining quantitative variables. Dietary information from the San Luis Valley population was used to estimate cholesterol intake identified. Allelic effects were estimated in these groups to gain insight into the effect of dietary cholesterol intake of the estimated allelic effects.

The study was renewed in fiscal year 1996 to determine the contribution of polymorphic variation in nine candidate genes involved in lipid metabolism [APO(a), APOD, hepatic lipase (HL), cholesteryl ester transfer protein (CETP), LDL receptor related protein (LRP), 3- hydroxy-3 methyl glutryl-coenzyme A (HMG COA), VLDL-receptor, Lecithin cholesterol acyletransferase (LCAT) and paraoxonase (PON)] in determining quantitative lipoprotein-lipid levels in Hispanics and non-Hispanic Whites of the San Luis Valley, Colorado. The study also determined the molecular basis of the functional mutation in the lipoprotein lipase (LPL) gene which is associated with plasma triglyceride and HDL cholesterol variations. The objectives were achieved by fulfilling the following specific aims: 1) by PCR, DNA sequencing and SSCP analyses, all coding exons and putative regulatory elements in the LPL gene of individuals who were homozygous for the HindIII restriction site to detect nucleotide changes in the coding region which affected directly triglycerides and HDL-cholesterol levels werescreened, in vitro mutagenesis and expression studies were conducted to confirm which of the putative functional mutations was the actual functional mutation; 2) genetic variations in genes coding for CETP, HL, LRP, APOD, HMG COA, VLDL-receptor, LCAT and PON were identified by PCR or standard Southern blotting techniques, and the impact of individual polymorphisms and the joint impact of polymorphisms at different loci (genotype-genotype interaction) in determining quantitative lipoprotein-lipid levels in Hispanics and non-Hispanic whites were estimated; and 3) the distribution of APO(a) kringle 4 and pentanucleotide polymorphisms were determined by SDS-agarose gel electrophoresis and PCR, respectively, and LP(a) levels were quantified by enzyme-linked immunosorbent assay, and the correlation between APO(a) polymorphisms and LP(a) levels were investigated.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-05; Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Kamboh — University of Pittsburgh

REFERENCES:
- [Background] Kamboh MI, Kelly LJ, Ahn YI, Ferrell RE. Genetic polymorphism of apolipoprotein A-IV in the chimpanzee: common deletion of a conserved 12-nucleotide tandem repeat. Hum Biol. 1994 Aug;66(4):625-38. PMID 8088751
- [Background] Rewers M, Kamboh MI, Hoag S, Shetterly SM, Ferrell RE, Hamman RF. ApoA-IV polymorphism associated with myocardial infarction in obese NIDDM patients. The San Luis Valley Diabetes Study. Diabetes. 1994 Dec;43(12):1485-9. doi: 10.2337/diab.43.12.1485. PMID 7958503
- [Background] Kamboh MI, Svitko CM, Williams ER, Ferrell RE, Pollitzer WS. Hypervariable polymorphism of APO(a) in blacks and whites as reflected by phenotyping. Chem Phys Lipids. 1994 Jan;67-68:283-92. doi: 10.1016/0009-3084(94)90148-1. PMID 8187225
- [Background] Ahn YI, Kamboh MI, Aston CE, Ferrell RE, Hamman RF. Role of common genetic polymorphisms in the LDL receptor gene in affecting plasma cholesterol levels in the general population. Arterioscler Thromb. 1994 May;14(5):663-70. doi: 10.1161/01.atv.14.5.663. PMID 8172843
- [Background] Kamboh MI, Friedlaender JS, Ahn YI, Ferrell RE. A common deletion polymorphism in the apolipoprotein A4 gene and its significance in lipid metabolism. Arterioscler Thromb. 1994 May;14(5):656-62. doi: 10.1161/01.atv.14.5.656. PMID 8172842
- [Background] Ahn YI, Ferrell RE, Hamman RF, Kamboh MI. Association of lipoprotein lipase gene variation with the physiological components of the insulin-resistance syndrome in the population of the San Luis Valley, Colorado. Diabetes Care. 1993 Nov;16(11):1502-6. doi: 10.2337/diacare.16.11.1502. PMID 7905375
- [Background] Cole SA, Aston CE, Hamman RF, Ferrell RE. Association of a PvuII RFLP at the lipoprotein lipase locus with fasting insulin levels in Hispanic men. Genet Epidemiol. 1993;10(3):177-88. doi: 10.1002/gepi.1370100304. PMID 8102341
- [Background] Ahn YI, Kamboh MI, Hamman RF, Cole SA, Ferrell RE. Two DNA polymorphisms in the lipoprotein lipase gene and their associations with factors related to cardiovascular disease. J Lipid Res. 1993 Mar;34(3):421-8. PMID 8096867
- [Background] Saha N, Kamboh MI, Ahn YA, Tay JS, Ferrell RE. Apolipoprotein H polymorphism and serum lipoprotein and apolipoprotein levels in two Asian populations. Ethn Dis. 1993 Summer;3(3):250-4. PMID 8167541
- [Background] Crews DE, Kamboh MI, Mancilha-Carvalho JJ, Kottke B. Population genetics of apolipoprotein A-4, E, and H polymorphisms in Yanomami Indians of northwestern Brazil: associations with lipids, lipoproteins, and carbohydrate metabolism. Hum Biol. 1993 Apr;65(2):211-24. PMID 8449482
- [Background] Sanghera DK, Aston CE, Saha N, Kamboh MI. DNA polymorphisms in two paraoxonase genes (PON1 and PON2) are associated with the risk of coronary heart disease. Am J Hum Genet. 1998 Jan;62(1):36-44. doi: 10.1086/301669. PMID 9443862
- [Background] Kamboh MI, Rewers M, Aston CE, Hamman RF. Plasma apolipoprotein A-I, apolipoprotein B, and lipoprotein(a) concentrations in normoglycemic Hispanics and non-Hispanic whites from the San Luis Valley, Colorado. Am J Epidemiol. 1997 Dec 15;146(12):1011-8. doi: 10.1093/oxfordjournals.aje.a009229. PMID 9420525
- [Background] Saha N, Wang G, Vasisht S, Kamboh MI. Influence of two apo A4 polymorphisms at codons 347 and 360 on non-fasting plasma lipoprotein-lipids and apolipoproteins in Asian Indians. Atherosclerosis. 1997 Jun;131(2):249-55. doi: 10.1016/s0021-9150(97)06112-1. PMID 9199279
- [Background] Sanghera DK, Saha N, Aston CE, Kamboh MI. Genetic polymorphism of paraoxonase and the risk of coronary heart disease. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1067-73. doi: 10.1161/01.atv.17.6.1067. PMID 9194756
- [Background] Kamboh MI, Aston CE, Nestlerode CM, McAllister AE, Hamman RF. Haplotype analysis of two APOA1/MspI polymorphisms in relation to plasma levels of apo A-I and HDL-cholesterol. Atherosclerosis. 1996 Dec 20;127(2):255-62. doi: 10.1016/s0021-9150(96)05966-7. PMID 9125316
- [Background] Harris M, Sanghera DK, Kamboh MI. Short report on DNA marker at candidate locus. Two new alleles in the tetranucleotide repeat polymorphism in the LDL-receptor-related protein (LRP) gene. Clin Genet. 1996 Jul;50(1):54-5. No abstract available. PMID 8891388
- [Background] Marshall JA, Kamboh MI, Bessesen DH, Hoag S, Hamman RF, Ferrell RE. Associations between dietary factors and serum lipids by apolipoprotein E polymorphism. Am J Clin Nutr. 1996 Jan;63(1):87-95. doi: 10.1093/ajcn/63.1.87. PMID 8604675
- [Background] Kamboh MI, Aston CE, Hamman RF. The relationship of APOE polymorphism and cholesterol levels in normoglycemic and diabetic subjects in a biethnic population from the San Luis Valley, Colorado. Atherosclerosis. 1995 Jan 20;112(2):145-59. doi: 10.1016/0021-9150(94)05409-c. PMID 7772075
- [Background] Mehdi H, Aston CE, Sanghera DK, Hamman RF, Kamboh MI. Genetic variation in the apolipoprotein H (beta2-glycoprotein I) gene affects plasma apolipoprotein H concentrations. Hum Genet. 1999 Jul-Aug;105(1-2):63-71. doi: 10.1007/s004399900089. PMID 10480357
- [Background] Chiu L, Hamman RF, Kamboh MI. Apolipoprotein A polymorphisms and plasma lipoprotein(a) concentrations in non-Hispanic Whites and Hispanics. Hum Biol. 2000 Oct;72(5):821-35. PMID 11126727
- [Background] Pfaff CL, Parra EJ, Bonilla C, Hiester K, McKeigue PM, Kamboh MI, Hutchinson RG, Ferrell RE, Boerwinkle E, Shriver MD. Population structure in admixed populations: effect of admixture dynamics on the pattern of linkage disequilibrium. Am J Hum Genet. 2001 Jan;68(1):198-207. doi: 10.1086/316935. Epub 2000 Dec 7. PMID 11112661
- [Background] Wang GQ, DiPietro M, Roeder K, Heng CK, Bunker CH, Hamman RF, Kamboh MI. Cladistic analysis of human apolipoprotein a4 polymorphisms in relation to quantitative plasma lipid risk factors of coronary heart disease. Ann Hum Genet. 2003 Mar;67(Pt 2):107-24. doi: 10.1046/j.1469-1809.2003.00023.x. PMID 12675687
- [Background] Razzaghi H, Day BW, McClure RJ, Kamboh MI. Structure-function analysis of D9N and N291S mutations in human lipoprotein lipase using molecular modelling. J Mol Graph Model. 2001;19(6):487-94, 587-90. doi: 10.1016/s1093-3263(00)00096-6. PMID 11552677
- [Background] Saha N, Aston CE, Low PS, Kamboh MI. Racial and genetic determinants of plasma factor XIII activity. Genet Epidemiol. 2000 Dec;19(4):440-55. doi: 10.1002/1098-2272(200012)19:43.0.CO;2-8. PMID 11108652
- [Background] Razzaghi H, Aston CE, Hamman RF, Kamboh MI. Genetic screening of the lipoprotein lipase gene for mutations associated with high triglyceride/low HDL-cholesterol levels. Hum Genet. 2000 Sep;107(3):257-67. doi: 10.1007/s004390000367. PMID 11071388
- [Background] Kamboh MI, Aston CE, Hamman RF. DNA sequence variation in human apolipoprotein C4 gene and its effect on plasma lipid profile. Atherosclerosis. 2000 Sep;152(1):193-201. doi: 10.1016/s0021-9150(99)00459-1. PMID 10996355